CLINICAL TRIAL: NCT04736875
Title: Study of the Hemodynamic and Clinical Maturation of the Native Arteriovenous Fistula for Hemodialysis
Brief Title: Arteriovenous Fistula Maturation Evaluation Study. FAME Study
Status: Completed | Type: Observational
Sponsor: Medifil AE (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Ioannis Emmanouel Giannikouris, Director Nephrologist, Medifil AE
Other Study IDs: 3
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: End-stage Renal Disease; Hemodialysis Access Failure; Vascular Access Maturation; Native Arteriovenous Fistula
Keywords: hemodialysis; native arteriovenous fistula; maturation; feeding artery; efferent vein
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dialysis: Patients with hemodialysis-dependent end-stage renal disease and a newly created native arteriovenous fistula
  Interventions: Diagnostic Test: Doppler ultrasound study

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound study — Transcutaneous Doppler ultrasound (DUS) study was performed at the mid brachial artery to assess diameter, VF and RI, and at the mid segment of the efferent vein to assess the diameter and wall thickness.

SUMMARY:
Study of the features of hemodynamic and clinical maturation of the native arteriovenous fistula for hemodialysis.

DETAILED DESCRIPTION:
This is a prospective, single-center, observational study, investigating the clinical and hemodynamic features of maturation of hemodialysis native arteriovenous fistula (AVF). Hemodynamic features under investigation are the diameter of the feeding brachial artery, volume of flow (VF) measured with transcutaneous Duplex ultrasound (DUS), resistivity index (RI), diameter and wall thickness of the efferent vein, measured at days 1, 2, 3, 4, 5, 6, 7, 14, 21, 30, 60 and 90 post creation. Clinical features of maturation are the time of first access successful cannulation and the performance of three consecutive adequate dialysis sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodialysis patients
2. new native arteriovenous fistula (AVF)

Exclusion Criteria:

1. Patients not eligible for AVF creation
2. Patients with non compensated heart failure New York Heart Association stages 3 and 4

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit patients with end-stage renal disease eligible for native arteriovenous fistula creation for hemodialysis fulfilling the study's inclusion critera.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Volume flow | day 1 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 2 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 3 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 4 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 5 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 6 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 7 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 14 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 21 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 28 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 60 post access creation
  Volume of flow in brachial artery in L/min
Volume flow | day 90 post access creation
  Volume of flow in brachial artery in L/min
brachial artery diameter | day 1 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 2 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 3 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 4 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 5 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 6 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 7 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 14 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 21 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 28 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 60 post access creation
  Diameter of the Brachial artery in mm
brachial artery diameter | day 90 post access creation
  Diameter of the Brachial artery in mm
Resistive index RI | day 1 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 2 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 3 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 4 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 5 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 6 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 7 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 14 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 21 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 28 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 60 post access creation
  Calculation of the Resistive Index of the Brachial artery
Resistive index RI | day 90 post access creation
  Calculation of the Resistive Index of the Brachial artery
Diameter of the efferent vein | day 1 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 2 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 3 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 4 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 5 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 6 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 7 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 14 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 21 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 28 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 60 post access creation
  Diameter of the the efferent vein in mm
Diameter of the efferent vein | day 90 post access creation
  Diameter of the the efferent vein in mm
Wall thickness of the efferent vein | day 1 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 2 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 3 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 4 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 5 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 6 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 7 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 14 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 21 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 28 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 60 post access creation
  Wall thickness of the efferent vein in mm
Wall thickness of the efferent vein | day 90 post access creation
  Wall thickness of the efferent vein in mm

SECONDARY OUTCOMES:
Time of first successful cannulation | 30 and 60 days
  Time period between access creation and first successful cannulation for hemodialysis
Successful hemodialysis | 30 and 60 days
  Three consecutive adequate hemodialysis sessions based on measurement of single pool kt/V
Primary patency | 6 months
  Percentage of total patent arteriovenous fistulae without the need of additional interventions assessed by transcutaneous dopler ultrasound
Surgeon-Nephrologist access site selection concordance | At access creation (day 0)
  Record of the opinion regarding the site of vascular access creation between the nephrologist performing preoperative mapping and the surgeon performing access creation with the use of a questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis E Giannikouris, MD, MSc, PhD, Principal Investigator — Mediterranean Hospital
Locations (1):
- Mediterranean Hospital, Glyfada, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided